CLINICAL TRIAL: NCT02360501
Title: Combination of Docetaxel, Cisplatin, and Capecitabine (DCX) in the Treatment of Locally Advanced or Metastatic Nasopharyngeal Carcinoma: a Prospective, Phase 2 Study
Brief Title: Combination of Docetaxel, Cisplatin, and Capecitabine (DCX) in the Treatment of Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liang Wang, Doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCX in NPC
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: nasopharyngeal carcinoma; induction chemotherapy; docetaxel; xeloda
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment arm (Experimental): docetaxel 75mg/㎡,d1; cisplatin 25mg/㎡,d1-3; capecitabine 2g/㎡, d1-14. repeated every three weeks
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — 75mg/㎡,d1
  Other Names: Taxotere
Drug: Cisplatin — 25mg/㎡,d1-3
Drug: Capecitabine — 2000mg/㎡,d1-14
  Other Names: xeloda

SUMMARY:
The standard treatment strategy for locally advanced (stage IVA) and metastatic (stage IVB) nasopharyngeal carcinoma has not been defined yet. Generally induction chemotherapy is given to those patients in order to shrink the tumor volume and facilitate the following radiation therapy. Thus, in this study, the investigators use the combination of Docetaxel+Cisplatin+Xeloda (DCX) to treat locally advanced and metastatic nasopharyngeal carcinoma patients, in order to evaluate the efficacy and safety profiles.

DETAILED DESCRIPTION:
The standard treatment strategy for locally advanced (stage IVA) and metastatic (stage IVB) nasopharyngeal carcinoma has not been defined yet. Generally induction chemotherapy is given to those patients in order to shrink the tumor volume and facilitate the following radiation therapy.However, the standard chemotherapy regimen has not been defined yet.Combination of cisplatin and fluracil is the commonly used regimen with tolerable toxicity. Recent studies have found that docetaxel has good efficacy on nasopharyngeal carcinoma patients, and capecitabine can be safely used instead of fluracil. Thus, in this study, we use the combination of Docetaxel+Cisplatin+Xeloda (DCX) to treat locally advanced and metastatic nasopharyngeal carcinoma patients, in order to evaluate the efficacy and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* stage IVA and IVB nasopharyngeal carcinoma
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.
* allergy to any of these three drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
overall response rate | every 4 weeks,up to completion of treatment(approximately 6 months)
  overall response rate is the sum of complete response rate and partial response rate.

SECONDARY OUTCOMES:
complete response rate | every 4 weeks,up to completion of treatment(approximately 6 months)
1 year progression free survival rate | date from diagnosis of NPC to disease progression, or death of any cause, whichever comes first （up to 12 months）.
1 year overall survival rate | date from diagnosis of NPC to death of any cause (up to 12 months)
safety profiles (including hematologic toxicities and non-hematologic toxicities.) | date from diagnosis of NPC to completion of study (about 6 months)
  including hematologic toxicities (eg.the incidence rate of neutropenia,thrombocytopenia, and anemia), and non-hematologic toxicities (eg.edema, diarrhea, hand-foot-syndrome).

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, DOCTOR, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China